CLINICAL TRIAL: NCT05423028
Title: The Effects of Vitamin B12 and Dextrose on the Ultrasound-guided Median Nerve Hydrodissection
Brief Title: Vitamin B12 and Dextrose for Median Nerve Hydrodissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCKUH-11103036
Record Dates: First submitted 2022-06-06; First posted 2022-06-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dextrose (Active Comparator)
  Interventions: Procedure: Ultrasound-guided nerve hydrodissection
- Vitamin B12 (Experimental)
  Interventions: Procedure: Ultrasound-guided nerve hydrodissection
- Dextrose + Vitamin B12 (Experimental)
  Interventions: Procedure: Ultrasound-guided nerve hydrodissection

INTERVENTIONS:
Procedure: Ultrasound-guided nerve hydrodissection — Peri- median nerve injection for hydrorelease and decompression

SUMMARY:
Carpal tunnel syndrome is the most common peripheral entrapment neuropathy of the upper limb. Previous experiments found that ultrasound-guided median nerve hydrodissection with 5% dextrose water could ameliorate the condition of carpal tunnel syndrome. Oral administration of vitamin B 12 had been reported to reduce the discomfort from peripheral neuropathy although the level of evidence is not strong. This prospective, double-blind randomized control trial aims to compare the effects of different kinds of the injection agents on carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis (carpal tunnel syndrome) was confirmed using an electrophysiological study.

Exclusion Criteria:

* Previously undergone wrist surgery or steroid injection for CTS
* Thrombocytopenia
* Coagulopathy
* Inflammation status
* Polyneuropathy
* Brachial plexopathy
* Cervical radiculopathy
* Autoimmune disease
* Malignancy
* Pregnancy

Thoracic outlet syndrome

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of Boston Carpal Tunnel Syndrome Questionnaire | Pre-treatment, 1st, 3rd, 6th month after injection
  Measure the severity of symptoms and functional status before and after treatment

SECONDARY OUTCOMES:
Visual analog scale of pain and tingling | Pre-treatment, 1st, 3rd, 6th month after injection
  Measure the pain and tingling scale before treatment and after treatment. (0 is for not at all pain/tingling, and 100 is for extremely pain/tingling.)
Cross-sectional area of the median nerve | Pre-treatment, 1st, 3rd, 6th month after injection
  Using the ultrasound to measure the cross-sectional area of the median nerve before and after treatment
Median nerve elastography | Pre-treatment, 1st, 3rd, 6th month after injection
  Using the ultrasound to measure the elastography of the median nerve before and after treatment
Median nerve conduction velocity and amplitude | Pre-treatment, 1st, 6th month after injection
  Antidromic sensory nerve conduction velocity and amplitude of the median nerve before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes